CLINICAL TRIAL: NCT02498548
Title: Eccentric Motor Control Training to Improve Human Spinal Cord Injury: Intervention for Hip and Knee Function
Brief Title: Training of Eccentric Lower Extremity Function After SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Notre Dame (Other)
Responsible Party: Principal Investigator, Michele Basso, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014H0386
Record Dates: First submitted 2015-07-09; First posted 2015-07-15 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Individuals with no spinal cord injury or other neurological deficits.
- Unexercised SCI Knee or Hip (No Intervention): Individuals with spinal cord injury who have been discharged from a locomotor training program at least 6 months prior to enrollment in this study. This group will serve as unexercised control for the "Trained SCI Knee" group or "trained SCI Hip" group
- Trained SCI Knee or Trained SCI Hip (Experimental): Individuals with spinal cord injury who have been discharged from a locomotor training program at least 6 months prior to enrollment in this study. Training will specifically focus on rehabilitation of the knee joint or the hip joint.
  Interventions: Behavioral: Trained SCI Knee or Trained SCI Hip

INTERVENTIONS:
Behavioral: Trained SCI Knee or Trained SCI Hip — Individuals with SCI will perform downhill walking training 3 times a week for 12 wks with a 4 wk follow-up period. This intervention will be delivered by trained therapists. In order to focus on rehabilitation of knee control or hip control, members of this group will be trained at slow to moderate gait speeds.
  Other Names: DH Knee; DH Hip
  Arms: Trained SCI Knee or Trained SCI Hip

SUMMARY:
This project will characterize lower extremity eccentric muscle function among individuals who have undergone locomotor training after spinal cord injury and will evaluate the effect of downhill training at moderate speeds - targeted to rehabilitation eccentric function of the knee or hip.

DETAILED DESCRIPTION:
Lower extremity eccentric motor control is is critically important for locomotor function but is impaired after spinal cord injury (SCI). Even after treadmill training, preliminary evidence indicates that eccentric deficits persist among individuals with SCI. This proposal aims to characterize eccentric motor control of the muscles about the knee or hip during locomotion and evaluate the efficacy of downhill gait training at moderate speeds as an intervention to improve eccentric function of the knee joint or hip joint during walking.

ELIGIBILITY:
Individuals with SCI:

Inclusion Criteria:

* medically approved
* discharged from outpatient rehabilitation for 6 months
* incomplete SCI based on ASIA impairment score (AIS C or D) at neurologic level C1-T10
* ability to take some steps overground and on the treadmill
* 18-90 years old.
* ability to speak English. Note: the quality of life measures have not been validated yet in non-English speaking populations.

Exclusion Criteria:

* evidence of lower motor neuron injury in the legs
* use of botox in the past 3 months
* pre-existing or confounding neurologic conditions (i.e. brain injury, stroke, HIV)
* acute deep vein thrombosis
* skin wounds in regions where harness or hands provide support
* pregnancy. Note: Persons who are pregnant will not be enrolled as exercise tolerance is unknown in these women with SCI.
* cognitive conditions that preclude providing informed consent
* ventilator-dependence as study results will be confounded by mobility limitations imposed by equipment
* persistent orthostatic hypotension (drop of BP >30mmHg in treadmill and harness equipment)
* hospitalization for myocardial infarction, cardiac surgery or congestive heart failure exacerbation within 3 months of enrollment in study
* participation in any other concurrent exercise programs.

Note: Use of anti-spasticity and other medications (dose, frequency) will be monitored throughout training and used as a confounding variable in the analyses.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-06; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in time to complete 6 minutes of level walking (i.e., the 6 minute walk test) | baseline, 12 weeks

SECONDARY OUTCOMES:
Change from baseline in time to complete 10 meters of level walking (i.e., the 10 meter walk test) | baseline, 12 weeks
Change from baseline in peak magnitude of sagittal knee power absorption or frontal Hip power during loading response | baseline, 12 weeks

OTHER OUTCOMES:
Change from baseline in maximum voluntary eccentric knee flexion contraction after performing eccentric activity on the contralateral limb (i.e., the contralateral priming effect) | baseline, 12 weeks
Change from baseline in Neuromuscular Recovery Scale score | baseline, 12 weeks
Change from baseline in balance function as measured by the Berg Balance Scale score | baseline, 12 weeks
Change from Baseline in SCI specific Quality of Life score | baseline, 12 weeks
Change from second baseline in time to complete 6 minutes of level walking (i.e., the 6 minute walk test) | 12 weeks, 16 weeks
Change from second baseline in time to complete 10 meters of level walking (i.e., the 10 meter walk test) | 12 weeks, 16 weeks
Change from second baseline in peak magnitude of sagittal knee power absorption or frontal hip power during loading response | 12 weeks, 16 weeks
Change from second baseline in maximum voluntary eccentric knee flexion contraction after performing eccentric activity on the contralateral limb (i.e., the contralateral priming effect) | 12 weeks, 16 weeks
Change from second baseline in Neuromuscular Recovery Scale score | 12 weeks, 16 weeks
Change from second baseline in balance function as measured by Berg Balance Scale score | 12 weeks, 16 weeks
Change from second baseline in SCI specific Quality of Life score | 12 weeks, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: D. Michele M Basso, Principal Investigator — Ohio State University
Locations (1):
- D Michele basso, Columbus, Ohio, United States